CLINICAL TRIAL: NCT04909125
Title: Standard Versus Investigatioinal Fractionation Trial - Nodal Radiation
Brief Title: Breast Fractionation Study - Standard Versus Investigational Fractionation Trial - Nodal Radiation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Collaborators: Northern Sydney and Central Coast Area Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SVIFT Nodal Trial
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Post Mastectomy
Keywords: radiotherapy; hypofractionation; quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Masking Description: Patients will be randomised to one of the arms and will be notified for the randomization results. Randomisation ratio 2:1 (hypofractionation : standard)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionation Arm (Active Comparator): 40Gy / 15 fractions, 2.67Gy per fraction, over 3.5 week (9 fractions per fortnight)
  Interventions: Radiation: Hypofractionated radiotherapy VS Standard/Conventional fractionation radiotherapy
- Standard /Conventional fractionation Arm (Other): 50Gy / 25 fractions, 2Gy per fraction, over 5.5 week (9 fractions per fortnight)
  Interventions: Radiation: Hypofractionated radiotherapy VS Standard/Conventional fractionation radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy VS Standard/Conventional fractionation radiotherapy — The purpose of this study is to investigate toxicity following standard conventional fractionation versus moderately hypofractionated radiotherapy to the breast, chest wall and regional lymph nodes

SUMMARY:
The purpose of this study is to investigate the difference in fatigue, quality of life and radiation morbidity between hypofractionated and conventional radiation to the breast, chest wall and regional lymph nodes post mastectomy or lumpectomy

DETAILED DESCRIPTION:
Breast cancer is the most commonly diagnosed cancer in Australia. Radiotherapy to the breast, chest wall and regional lymph nodes for breast cancer after surgery can reduce the risk of local recurrence by 50% and reduce breast cancer mortality. Traditionally, radiotherapy is delivered in a large number of small doses i.e. 25 treatment sessions over 5 1/2 weeks. Another approach is to give a lower number of larger doses i.e. 15 sessions over 3 1/2 weeks (hypofractionated radiotherapy).

Several studies in Europe and Asia have investigated hypofractionated radiotherapy to the chest wall, breast and regional lymph nodes following surgery for breast cancer, and found that it is equally effective to standard treatment, with similar side effects. These two approaches have not been directly compared in Australia.

This trial is to compare these two approaches, to determine whether hypofractionated radiotherapy is better tolerated by patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* ECOG performance status 0-2
* Ability to understand and willingness to sign a written informed consent document
* Stage pT1-3, pN0-3, M0 histologically proven breast cancer no matter the status of ER/PR/HER2 receptor testing
* Managed with either mastectomy or breast conserving surgery
* Suitable for radiation therapy to the breast/chest wall and regional lymph nodes
* Neoadjuvant and adjuvant systemic therapy with chemotherapy, endocrine therapy and anti-HER2 therapy is accepted
* Neoadjuvant radiotherapy (reverse sequencing) accepted
* Breast implants and expanders are accepted
* Patients with connective tissue disease are allowed if the treating radiation oncologist finds radiation therapy indicated
* Life expectancy minimum 10 years
* Patients with non-breast malignancies are accepted if the patient has been disease free for five years and/or has a low risk of recurrence as estimated by the treating radiation oncologist (to be determined at initial patient appointment)

Exclusion Criteria:

* Prior radiotherapy to the ipsilateral breast or chest wall
* Pregnancy or lactation
* Radiosensitivity syndrome
* Permanent pacemaker/defibrillator within radiotherapy field
* Oncoplastic surgery where boost volume unacceptable (clinician discretion)
* Conditions indicating that the patient cannot go through radiation therapy or follow up, or a condition where the treating oncologist thinks the patient should not participate in the trial (for example, language barriers)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue | six weeks post radiation treatment
  Changes in patient reported fatigue at six weeks post commencing radiotherapy compared to baseline fatigue score. Fatigue score is rated as fatigue that interfered with patients' normal daily activities from "all of the time", "most of the time", "a good bit of the time", "some of the time", "a little of the time", "hardly any of the time", "none of the time" with the "all of the time" being the worst outcome

SECONDARY OUTCOMES:
Changes in patients' quality of life | first to 8th weeks post radiation treatment, half yearly for 2 years, annually for 3 years
  Changes in patients' quality of life during radiotherapy and follow up period are captured by questionnaires. The questions are for examples how difficult is it in planning or being able to continue your usual activities?, how often have you felt low in energy? The score scales are from "all of the time", "most of the time", "a good bit of the time", "some of the time", "a little of the time", "hardly any of the time", "none of the time" with the "all of the time" being the worst outcome
Number of participants with acute radiation dermatitis in irradiated area | During treatment
  Grade 2 or worse radiation dermatitis
Number of participants with ipsilateral arm lymphoedema | 3 years post radiation treatment
  The circumference of the ipsilateral arm >=10% increased compared to the other arm defines oedema
Number of participants with ipsilateral arm range of motion | 3 years post radiation treatment
  Impaired shoulder movement is present when >20 degrees difference between arms at flexion and/or abduction
Disease Recurrence | 5 years from treatment
  Any disease progression or recurrence - location and time of event
Self reported acute & late radiation toxicities | first to 8th weeks post radiation treatment, half yearly for 2 years, annually for 3 years
  acute radiation toxicities during treatment and late radiation toxicities are captured by questionnaires
Compare the indirect radiation therapy costs by 2 treatment arms | 4 weeks post radiation treatment
  data of cost of attending treatment, work and lifestyle impact are captured by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Susan Carroll, MBBS FRANZCR, Principal Investigator — Radiation Oncology Department, Royal North Shore Hospital
Locations (1):
- Radiation Oncology, Northern Sydney Cancer Centre, Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No